CLINICAL TRIAL: NCT03514823
Title: Respiratory Muscle Contribution to Blood Pressure During Exercise in Healthy Humans
Brief Title: Respiratory Muscle Contribution to Blood Pressure During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Thomas P. Olson, M.S., Ph.D., Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-011100; 5R01HL126638-03 (NIH)
Record Dates: First submitted 2018-04-18; First posted 2018-05-02 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Respiratory Muscle; Blood Pressure; Exercise Capacity; Sympathetic Nerve Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT Group (Experimental)
  Interventions: Other: Inspiratory Muscle Training (IMT)
- No IMT Group (Sham Comparator)
  Interventions: Other: No Inspiratory Muscle Training (IMT)

INTERVENTIONS:
Other: Inspiratory Muscle Training (IMT) — Inspiratory muscle training (IMT) are breathing exercises used to increase strength and endurance of the respiratory muscles.
  Arms: IMT Group
Other: No Inspiratory Muscle Training (IMT) — No inspiratory muscle training.
  Arms: No IMT Group

SUMMARY:
The investigators seek to understand how reflexes from the breathing muscles influence blood pressure during exercise. Furthermore, the investigators are determining if increasing breathing muscle strength (via inspiratory muscle training) influences the respiratory muscle contribution to blood pressure during exercise.

ELIGIBILITY:
Healthy participants with no history of cardiovascular, pulmonary, neurologic, orthopedic or other neuromuscular diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
VO2 max test | Through study completion, an average of one year.
  Using a MedGraphics metabolic cart, the investigators will measure the maximum amount of oxygen that an individual can utilize during exercise. During this test the subject will be asked to exercise to his/her max capacity on a recumbent bicycle while breathing through a mouth piece that is hooked into the MedGraphics computer software.
Blood Pressure | Through study completion, an average of one year.
  Blood pressure will be taken every few minutes during exercise testing using a standard blood pressure cuff to monitor changes in blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Olson, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials